CLINICAL TRIAL: NCT02834637
Title: A Dose Reduction Immunobridging and Safety Study of Two HPV Vaccines in Tanzanian Girls
Acronym: DoRIS
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: University of York (Other); Institut Català d'Oncologia (Other); National Cancer Institute (NCI) (NIH); Karolinska Institutet (Other); Technische Universität Berlin (Other); Tanzanian National Institute for Medical Research (Unknown); University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MITU-002
Record Dates: First submitted 2016-06-29; First posted 2016-07-15 (Estimated); Last update posted 2025-09-10 (Actual); Status verified 2025-03

CONDITIONS: Human Papilloma Virus
Keywords: HPV; cervical cancer; vaccines; HPV vaccine; dose reduction; Human papilloma virus vaccine schedules
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — human papillomavirus vaccine, L1 type 16, 18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- 3 doses 2valent (Active Comparator): 3 doses of bivalent HPV vaccine (Cervarix) given at M0, M1 and M6
  Interventions: Drug: bivalent HPV vaccine
- 2 doses 2valent (Active Comparator): 2 doses of bivalent HPV vaccine (Cervarix) given at M0 and M6
  Interventions: Drug: bivalent HPV vaccine
- 1 dose 2valent (Active Comparator): 1 dose of bivalent HPV vaccine (Cervarix) given at M0
  Interventions: Drug: bivalent HPV vaccine
- 3 doses 9valent (Active Comparator): 3 doses of nonavalent HPV vaccine (Gardasil9) given at M0, M2 and M6
  Interventions: Drug: nonavalent HPV vaccine
- 2 doses 9valent (Active Comparator): 2 doses of nonavalent HPV vaccine (Gardasil9) given at M0 and M6
  Interventions: Drug: nonavalent HPV vaccine
- 1 dose 9valent (Active Comparator): 1 dose of nonavalent HPV vaccine (Gardasil9) given at M0
  Interventions: Drug: nonavalent HPV vaccine

INTERVENTIONS:
Drug: bivalent HPV vaccine — head to head comparisons of different dose schedules and HPV vaccine types
  Other Names: Cervarix
  Arms: 1 dose 2valent; 2 doses 2valent; 3 doses 2valent
Drug: nonavalent HPV vaccine — head to head comparisons of different dose schedules and HPV vaccine types
  Other Names: Gardasil9
  Arms: 1 dose 9valent; 2 doses 9valent; 3 doses 9valent

SUMMARY:
Cervical cancer is the most common cancer in women aged 15-44 years in East Africa, and mortality rates are very high. HPV vaccines are most effective if given to girls who have not yet acquired HPV infection. In Tanzania, HPV vaccine has been shown to be safe, acceptable and can be delivered with high coverage (~80%). However, the cost of delivering HPV vaccine is considerably higher than costs for traditional infant/child vaccinations. This is primarily because of costs to establish outreach programmes and associated personnel costs including nurses who must spend significant time away from their posts to deliver vaccine, especially if multiple doses are needed. There is global interest in simplifying HPV vaccine delivery by reducing the number of doses. If a single dose could be given, this could halve the costs of delivery, making it more accessible to the populations that need it most. Recently, the WHO recommended that 2 doses of HPV vaccine could be given to young girls, based on studies in high and upper middle-income countries. However in Africa high rates of infections like malaria and worms can affect immune responses to vaccines. It is essential to know that reducing the number of doses does not reduce the protective immune response of these vaccines. The investigators are conducting a trial in Tanzanian girls aged 9-14 years to establish whether a single dose of HPV vaccine produces immune responses that are likely to be effective in preventing cervical cancer. Two different HPV vaccines, the bivalent (2-v) vaccine that protects against HPV 16/18 (the cause of 70% of cancers) and the 9-valent (9-v) vaccine that protects against 9 HPV types, will be compared. The trial will randomise 900 girls to 6 arms and follow them for 36 months. Girls will receive the 2-v or the 9-v HPV vaccine, as 1, 2 or 3 doses. Girls receiving 1 or 2 doses will be compared with those receiving 3 doses of the same vaccine, to ensure that the reduced dose regimen produces an immune response that is not inferior to 3 doses. Girls in the 1 and 2 dose arms will be enrolled in an extension and followed for up to 9 years, to examine the stability of immune responses. The immune responses in this study will also be compared with results from other countries where the vaccine has been shown to be protective. This will provide information about whether a reduced number of doses is likely to be protective in Africa. This work will be extremely important in informing future HPV vaccination strategies and will be one of the first randomised trials of 1 and 2 doses of any HPV vaccine in Africa.

DETAILED DESCRIPTION:
Human papillomavirus (HPV) infection is the primary cause of cervical cancer, a major public health problem in Africa. Currently there are three vaccines (Cervarix, Gardasil® and Gardasil-9®) that offer excellent protection against HPV infection with vaccine-related HPV genotypes. The objective of this trial is to demonstrate non-inferiority of immune responses with 1 dose of HPV vaccine compared with the recommended 2 or 3 doses of the same vaccine by evaluating HPV 16/18-specific seropositivity, antibody avidity and memory B cell responses at M36. Specifically, the investigators will determine whether a single dose of the 2-valent HPV vaccine (Cervarix, that protects against HPV 16/18 genotypes) or of a new 9-valent HPV vaccine (Gardasil-9,that protects against HPV 6/11/16/18/31/33/45/52/58) produces immune responses that are non-inferior to those observed with 3 doses of vaccine when given to HIV-negative 9-14 years old girls in a malaria-endemic region of Tanzania.

The trial will also determine whether the World Health Organization's (WHO) recently recommended 2 dose strategy for girls aged under 15 years produces similar immune responses in Sub-Saharan Africa (SSA) compared to the previously recommended 3 dose schedule. In addition, the cost-effectiveness of alternative dosing schedules and of the two vaccines will be explored.

The trial will enrol 900 girls who are resident in Mwanza into an un-blinded, individually-randomised trial with 6 arms. Arm A will comprise participants randomised to receive 3 doses of the 2-valent vaccine, Arm B those randomised to receive 2 doses of the 2-valent vaccine and Arm C those randomised to receive 1 dose of the 2-valent vaccine. Arms D, E and F will be those participants randomised to receive 3, 2 or 1 dose of the 9-valent vaccine, respectively.

The effect of different dose schedules and type of HPV vaccine on a range of immune responses will be measured up to 36 months after the first dose. In a trial extension that will extend follow-up, we will also determine whether the one dose schedule of these vaccines produces non-inferior immune responses to the recommended two dose schedule for up to 108 months, and examine the long-term stability of the immune responses to 9 years after the first dose.

The protocol will be harmonised, and laboratory procedures and immunological endpoints will be cross-validated, with those of a large HPV vaccine dose-reduction efficacy trial being planned by the NIH in Costa Rica to examine the protective effect of the same vaccines given as 1 or 2 doses. This trial will allow the examination of quality and durability of antibody responses, and safety and cost-effectiveness of reduced dose schedules compared to the originally recommended 3 dose schedule in a population with high burden of malaria and other infections that may affect vaccine immune responses.

ELIGIBILITY:
Inclusion Criteria:

* Born female;
* Aged between 9 and 14 years inclusive;
* Enrolled in a government primary or secondary day school in Mwanza city (or neighbouring district if included);
* Living in Mwanza city (or neighbouring district if included) without plans to move away in the next 36 months;
* Willing to participate in the study and sign the informed assent form;
* Supported in this study participation by at least one of their parents (or LAR), who has signed the informed consent document;
* In good health as determined by a medical history (a physical examination will be conducted if necessary according to the clinician's judgement); and
* Able to pass a Test of Understanding (TOU) if aged 12 years or above, or if younger than 12 years old, a parent or LAR is able to pass a TOU

Exclusion Criteria:

* They are diagnosed with chronic conditions, such as autoimmune conditions, degenerative diseases, neurologic or genetic diseases among others;

  * They are HIV positive, or immunocompromised;
  * They are pregnant, less than three months post-partum or currently breastfeeding;
  * They are allergic to one of the vaccine components or to latex;
  * They are sexually active and are not willing to use an effective birth control method from 28 days before the first dose until 60 days after the last vaccine dose;
  * The nurse or clinician determining the eligibility, in agreement with principal investigator, considers that there is a reason that precludes participation;
  * They have been previously vaccinated against HPV

Ages: 9 Years to 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 930 (Actual)
Dates: Start 2017-02-23 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
non-inferiority of antibody seropositivity of 1 dose compared with 2 or 3 doses of the same vaccine | Month 24
  Proportion with HPV 16/18-specific seropositivity
non-inferiority of antibody geometric mean titre (GMT) of 1 dose of either vaccine compared with historical cohorts of women who received 1 dose in whom efficacy has been demonstrated | Month 24
  Geometric mean HPV 16/18 titre
non-inferiority of antibody seropositivity of 1 dose compared with 2 doses of the same vaccine | Month 60 and Month 108
  Proportion with HPV 16/18-specific seropositivity

SECONDARY OUTCOMES:
non-inferiority of HPV 16/18 seropositivity after 1 dose compared with 2 or 3 doses of the same vaccine | Month 12 and Month 36
  Proportion with HPV 16/18-specific seropositivity
evaluate HPV 16/18 seropositivity and antibody GMT at all time points when comparing 2 doses with 3 doses of the same vaccine. | Month 7, Month 12, Month 24 and Month 36
  HPV 16/18-specific seropositivity and antibody GMT
equivalence of HPV 16/18 seropositivity and antibody GMT at all time points when comparing the same dose regimen between the 2 vaccine types | Month 12, Month 24, Month 36, Month 60, Month 84 and Month 108
  HPV 16/18-specific seropositivity and antibody GMT
evaluate HPV 16/18 antibody avidity and memory B cell responses at all time points, comparing different dose regimens of the same vaccine and the same dose regimen between the two vaccines | Month 12, Month 24, Month 36, Month 84 and Month 108 (avidity); Month 12, Month 24 and Month 36 (memory B cells)
  HPV 16/18-specific antibody avidity and memory B cell responses
stability of antibody responses when comparing within the same arm. | Month 36, Month 60 and M108
  HPV 16/18-specific antibody GMT
evaluate HPV 16/18 seropositivity when comparing 1 dose of either vaccine with historical cohorts of women who received 1, 2 or 3 doses, in whom efficacy has been demonstrated | Month 24
  HPV 16/18-specific seropositivity
evaluate HPV 16/18 seropositivity when comparing the 2 dose regimen of either vaccine with historical cohorts of women who received 3 doses, in whom efficacy has been demonstrated | Month 24
  HPV 16/18-specific seropositivity
non-inferiority of HPV 16/18 antibody GMT when comparing the 2 dose regimen of either vaccine with historical cohorts of women who received 3 doses, in whom efficacy has been demonstrated | Month 24
  HPV 16/18-specific antibody GMT
evaluate HPV 6/11/31/33/45/52/58 antibody seropositivity with the 1 and 2 dose regimens of the 9-valent vaccine compared with the 3-dose regimen | Month 12, Month 24 and Month 36
  HPV 6/11/31/33/45/52/58-specific antibody seropositivity
evaluate HPV 6/11/31/33/45/52/58 antibody GMT with the 1 and 2 dose regimens of the 9-valent vaccine compared with the 3-dose regimen | Month 12, Month 24 and Month 36
  HPV 6/11/31/33/45/52/58-specific antibody GMT
unit cost of 1 dose regimens compared with 2 and 3 dose regimens | up to Month 36
  incremental financial and economic costs of vaccination, using WHO costing tool
cost-effectiveness of 1 dose regimens compared with 2 and 3 dose regimens, and of the 9-valent vaccine compared with the 2-valent vaccine | up to Month 36
  estimates of costs and effects of vaccination will be integrated into an existing HPV cost-effectiveness model (WHO CHOICE)
number of participants with treatment related solicited adverse events | within 30 days after each dose
  solicited adverse events considered to have a reasonable possibility of having been contributed to by the vaccine
number of participants with treatment related unsolicited adverse events | up to Month 36
  unsolicited adverse events considered to have a reasonable possibility of having been contributed to by the vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Watson-Jones, Dr, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Mwanza Intervention Trials Unit (MITU), Mwanza, Tanzania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Baisley K, Kemp TJ, Kreimer AR, Basu P, Changalucha J, Hildesheim A, Porras C, Whitworth H, Herrero R, Lacey CJ, Schiller JT, Lucas E, Mutani P, Dillner J, Indangasi J, Muwonge R, Hayes RJ, Pinto LA, Watson-Jones D. Comparing one dose of HPV vaccine in girls aged 9-14 years in Tanzania (DoRIS) with one dose of HPV vaccine in historical cohorts: an immunobridging analysis of a randomised controlled trial. Lancet Glob Health. 2022 Oct;10(10):e1485-e1493. doi: 10.1016/S2214-109X(22)00306-0. PMID 36113532
- [Background] Baisley KJ, Whitworth HS, Changalucha J, Pinto L, Dillner J, Kapiga S, de Sanjose S, Mayaud P, Hayes RJ, Lacey CJ, Watson-Jones D. A dose-reduction HPV vaccine immunobridging trial of two HPV vaccines among adolescent girls in Tanzania (the DoRIS trial) - Study protocol for a randomised controlled trial. Contemp Clin Trials. 2021 Feb;101:106266. doi: 10.1016/j.cct.2021.106266. Epub 2021 Jan 6. PMID 33421649
- [Background] Watson-Jones D, Changalucha J, Whitworth H, Pinto L, Mutani P, Indangasi J, Kemp T, Hashim R, Kamala B, Wiggins R, Songoro T, Connor N, Mbwanji G, Pavon MA, Lowe B, Mmbando D, Kapiga S, Mayaud P, de SanJose S, Dillner J, Hayes RJ, Lacey CJ, Baisley K. Immunogenicity and safety of one-dose human papillomavirus vaccine compared with two or three doses in Tanzanian girls (DoRIS): an open-label, randomised, non-inferiority trial. Lancet Glob Health. 2022 Oct;10(10):e1473-e1484. doi: 10.1016/S2214-109X(22)00309-6. PMID 36113531
- [Background] Watson-Jones D, Changalucha J, Maxwell C, Whitworth H, Mutani P, Kemp TJ, Kamala B, Indangasi J, Constantine G, Hashim R, Mwanzalima D, Wiggins R, Mmbando D, Connor N, Pavon MA, Lowe B, Kapiga S, Mayaud P, de Sanjose S, Dillner J, Hayes RJ, Lacey CJ, Pinto L, Baisley K. Durability of immunogenicity at 5 years after a single dose of human papillomavirus vaccine compared with two doses in Tanzanian girls aged 9-14 years: results of the long-term extension of the DoRIS randomised trial. Lancet Glob Health. 2025 Feb;13(2):e319-e328. doi: 10.1016/S2214-109X(24)00477-7. PMID 39890232
- [Background] Baisley K, Kemp TJ, Mugo NR, Whitworth H, Onono MA, Njoroge B, Indangasi J, Bukusi EA, Prabhu PR, Mutani P, Galloway DA, Mwanzalime D, Kapiga S, Lacey CJ, Hayes RJ, Changalucha J, Pinto LA, Barnabas RV, Watson-Jones D. Comparing one dose of HPV vaccine in girls aged 9-14 years in Tanzania (DoRIS) with one dose in young women aged 15-20 years in Kenya (KEN SHE): an immunobridging analysis of randomised controlled trials. Lancet Glob Health. 2024 Mar;12(3):e491-e499. doi: 10.1016/S2214-109X(23)00586-7. PMID 38365419
- [Derived] Kemp TJ, Baisley K, Changalucha J, Indangasi J, Whitworth H, Lacey CJ, Mwanzalima D, Hashim R, Kapiga S, Hayes RJ, Pinto LA, Watson-Jones D. Immunogenicity of one and two doses of Gardasil(R)9 in Tanzanian girls in the DoRIS Trial. NPJ Vaccines. 2025 Dec 19. doi: 10.1038/s41541-025-01344-1. Online ahead of print. PMID 41419735
- [Derived] Hsiao A, Struckmann V, Stephani V, Mmbando D, Changalucha J, Baisley K, Levin A, Morgan W, Hutubessy R, Watson-Jones D, Whitworth H, Quentin W. Costs of delivering human papillomavirus vaccination using a one- or two-dose strategy in Tanzania. Vaccine. 2023 Jan 9;41(2):372-379. doi: 10.1016/j.vaccine.2022.11.032. Epub 2022 Nov 29. PMID 36460537